CLINICAL TRIAL: NCT06951230
Title: The Efficacy of Scalp Block Versus Intravenous Fentanyl in Pain Control Intraoperatively in Craniotomy Patients
Brief Title: The Efficacy of Scalp Block in Craniotomy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: FMASU MS72/2024
Record Dates: First submitted 2025-04-04; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-02

CONDITIONS: Post-operative Pain; Narcotics Consumption; Pain Assessment; Intraoperative Hemodynamic Instability
Keywords: scalp block; pain; craniotomy; Pain control
MeSH Terms: conditions — Pain, Postoperative; Pain; Agnosia | interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- fentanyl group (Active Comparator): patients will receive general anesthesia followed by intravenous fentanyl (1ug/kg/hr)
  Interventions: Drug: Fentanyl injection
- scalp block group (Active Comparator): patients will receive general anesthesia followed by the scalp block.
  Interventions: Drug: Fentanyl injection; Procedure: scalp block

INTERVENTIONS:
Drug: Fentanyl injection — Fentanyl 1mcg/kg will be given before skin incision and Mayfield placement and followed up by fentanyl 1mcg/kg/hr, along the operation.
Procedure: scalp block — The scalp block procedure is performed with the patient in the supine position, utilizing surface landmarks for guidance. The local anesthetic is injected into the nerves after careful aspiration and under strict aseptic technique. The nerves that are typically injected include the supraorbital, supratrochlear, zygomaticotemporal, auriculotemporal, as well as the lesser and greater occipital nerves, with or without the inclusion of the third occipital nerve. The volume of 0.5% bupivacaine injected should not exceed 2 ml at each site.
  Arms: scalp block group

SUMMARY:
The aim of the study is to compare the effectiveness and safety of scalp block versus intravenous fentanyl in pain control intraoperatively in craniotomy patients. Most of the previous studies compared the effect of scalp block versus fentanyl or opioids in postoperative pain

DETAILED DESCRIPTION:
The history will be obtained from patient. The patients fasting 8 hours preoperatively will be examined and assessed, especially neurologically, to exclude any neurological deficit that may affect the results. Pre-operative laboratories will be reviewed for all patients as (complete blood picture, renal function tests, liver function tests, and coagulation profile) .

Patients will be assigned randomly by using a computer -generated table of random numbers, placing them in sealed envelopes, into two groups:

* Group A: (n= 10): patients will receive general anesthesia followed by intravenous fentanyl (1ug/kg/hr)
* Group B (control group): (n= 10): patients will receive general anesthesia then receive scalp block In the operating room, the monitor will be connected to track pulse oximetry (SpO2), non-invasive blood pressure (NIBP), and heart rate (HR). A second recording will occur after induction. An IV cannula will be inserted, and an electrocardiogram (ECG) obtained.

Pre-oxygenation with 100% oxygen will last 3 minutes, followed by IV induction with Propofol (2 mg/kg), Atracurium (0.5 mg/kg), and Fentanyl (1 mcg/kg). The patient will be placed on inhaled Isoflurane, and smooth intubation will be performed. Invasive blood pressure monitoring will be set up via the non-dominant radial artery, and a central venous line will be inserted in the internal jugular vein using ultrasound.

A scalp block will be done blindly for group B, while group A will receive Fentanyl (1 mcg/kg/hr) prior to Mayfield placement and skin incision. Throughout the operation, continuous monitoring of Electrocardiogram, Heart rate, invasive blood pressure (IBP), oxygen saturation and urine output will occur.

The scalp block will be performed under aseptic conditions by qualified personnel, with the patient in the supine position, using a landmark technique to target the relevant nerves for the blockage in group A.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 60
* Physical status: ASA I and II
* Elective operation, under general anaesthesia,

Exclusion Criteria:

* ASA above ll
* Patients with known uncontrolled comorbidities such as hypertension or Diabetes Mellites
* Coagulopathy, use of anti-coagulant or anti-platelet therapy.
* Known allergies to drugs used (Bupivacaine)
* Infection at the site of injection
* History of cranial nerve affection
* Emergency craniotomy.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
intra-operative hemodynamic stability | intra-operatively
  Recording the mean arterial blood pressure and heart rate readings will be obtained before induction , on skin pinning, on skin incision , 1 hour post induction, after 2hours and every hour hour till the end of the surgery

SECONDARY OUTCOMES:
fentanyl consumption | intra-operatively
  The total amount of fentanyl required along the operation will be recorded to detect the effect of the scalp block on narcotic consumption.

OTHER OUTCOMES:
post-operative pain | 1 hour post-operatively
  The pain is assessed post operatively in all patients 1 hour post-operatively using visual analogue scale a scale from 0 to 10 , where 0 is no pain and 10 is the worst unbearable pain. the amount of opiods needed will be recorded to detect the effect of the scalp block on postoperative pain control and decreasing narcotic demand.

CONTACTS AND LOCATIONS:
Overall Officials: Hegazy, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All dana will be shared once study is completed
Supporting Information: Study Protocol, SAP, ICF
Time Frame: before 6/2025
Access Criteria: free